CLINICAL TRIAL: NCT03137940
Title: A Study on Safety and Feasibility of a Session of Transcranial Electrical Stimulation (tDCS "One-shot") in Children and Young Adults With Unilateral Cerebral Palsy (UCP)
Brief Title: A Study on Safety of tDCS One-shot in UCP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Fondazione Stella Maris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: Safety_tDCS1.0
Record Dates: First submitted 2017-04-18; First posted 2017-05-03 (Actual); Last update posted 2019-08-08 (Actual); Status verified 2019-08

CONDITIONS: Hemiplegic Cerebral Palsy
Keywords: Unilateral Cerebral Palsy; tDCS; Safety; Upper Limb functions

STUDY DESIGN:
Intervention Model Description: Each subject receives, randomly, a real session of tDCS and a sham session with BrainStim Stimulator.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The medical device randomly assigns, to each subject, the sequence of the type of sessions, so no one knows the kind of session performed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- real tDCS (Experimental): one-shot of real tDCS session (1.5mA; 0.06 mA/cm2 for 20 minutes) with BrainStim Stimulator. The anode electrode is placed in a primary motor cortex (M1) of ipsilesional hemisphere (EEG 10/20 system), while cathode is placed in the supraorbital region (SO) of the contralateral hemisphere.
  Interventions: Device: real tDCS
- Sham tDCS (Sham Comparator): one-shot of sham tDCS session with BrainStim Stimulator (20 minutes). The montage of the electrodes will be placed as in the experimental session i.e.the anode electrode will be placed in a primary motor cortex (M1) of ipsilesional hemisphere (EEG 10/20 system), while cathode in the supraorbital region (SO) of the contralateral hemisphere.
  Interventions: Device: sham tDCS

INTERVENTIONS:
Device: real tDCS — one-shot of real tDCS session (1.5mA; 0.06 mA/cm2 for 20 minutes) with BrainStim Stimulator.
  Arms: real tDCS
Device: sham tDCS — one-shot of sham tDCS session (20 minutes) with BrainStim Stimulator.
  Arms: Sham tDCS

SUMMARY:
The study aims to evaluate the safety and the feasibility of transcranial Direct Current Stimulation (tDCS) session in children and young adults with Unilateral Cerebral Palsy (UCP). Secondarily it aims to test the effects of tDCS (real vs sham) in improving, in very short term, Upper Limb (UL) functions.

DETAILED DESCRIPTION:
Unilateral Cerebral Palsy (UCP) represents the most frequent form of CP; the upper limb (UL) is generally more affected than the lower limb with an impact in "activity" and "participation" areas. The non-invasive brain stimulation techniques (NIBS), such as transcranial Direct Current Stimulation (tDCS), appear able to modulate neuronal plasticity processes even more late in age attracting great interest for their potential fallout in the field of rehabilitation. The effects of tDCS in recovery of motor function has more investigated in adults, while in the pediatric population studies on safety and efficacy are still few and not conclusive. This study aims to evaluate the safety and the feasibility of tDCS session in children and young adults with UCP both in short term and in follow up (up to 24 hrs after the tDCS session). Secondarily it aims to test the effects of tDCS (real vs sham) in improving, in short term, UL functions. For the study 6 children (aged 10-17 years) and 6 young adults (aged 18-28 years) with UCP will be recruited. Each subject receives, randomly, a real session and a sham session of tDCS with BrainStim Stimulator. Before (T0), immediately after (T1) and after 1 hour and half (T2) to each tDCS session (real or sham) heart rate, blood pressure and UL functions will be measured. Moreover the subject fills in an ad hoc questionnaire on safety at T1 and T2 and, on call, at 24 hours after the sessions (T3).

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic Unilateral Cerebral Palsy
* Informed consent

Exclusion Criteria:

* Any contraindication for tDCS

Ages: 10 Years to 28 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 8 (Actual)
Dates: Start 2017-03-20 (Actual); Primary Completion 2017-10-20 (Actual); Study Completion 2017-12-30 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment Emergent Adverse Events [Safety and Tolerability] | The questionnaire will be filled in immediately after the tDCS session (T1), at 1 hour and half from T1 (T2) and, on call, at 24 hours from the tDCS session (T3)
  An adapted and child-friendly safety and tolerability questionnaire will be used for children and adolescent, while for young adults a questionnaire already used for this evaluation will be proposed. To explore the long-term safety the questionnaire is enriched with questions about quality of sleep, mood and activities to be answered after 24 hours of tDCS session

SECONDARY OUTCOMES:
Changes in heart rate [heartbeats per minute] | At baseline (T0, before the tDCS session), immediately after the tDCS session (i.e. 20 minutes after T0), at 1 hour and half from T1 (T2)
  The heart rate will be measured with an electronic device.
Changes in blood pressure [mmHg] | At baseline (T0, before the tDCS session), immediately after the tDCS session (i.e. 20 minutes after T0), at 1 hour and half from T1 (T2)
  The blood pressure will be measured with an electronic device.
Changes in Box and Block Test (BBT) | At baseline (T0, before the tDCS session), immediately after the tDCS session (i.e. 20 minutes after T0), at 1 hour and half from T1 (T2)
  The BBT measures unilateral gross-manual dexterity; subjects have to move, one by one, the maximum number of blocks from one compartment of a box to another within 60 seconds. The test will be performed firstly with the dominant hand and after with the contralateral. The patient is allowed a 15-second trial period prior to testing. ICF Domain: Activity
Changes in Hand Grip | At baseline (T0, before the tDCS session), immediately after the tDCS session (i.e. 20 minutes after T0), at 1 hour and half from T1 (T2)
  The hand grip will be measured with a dynamometer. The measurement will be performed firstly with the dominant hand and after with the contralateral.

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Cioni, MD, Study Director — IRCCS Fondazione Stella Maris, Università di Pisa
Locations (1):
- IRCCS Fondazione Stella Maris, Calambrone, Pisa, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Inguaggiato E, Bolognini N, Fiori S, Cioni G. Transcranial Direct Current Stimulation (tDCS) in Unilateral Cerebral Palsy: A Pilot Study of Motor Effect. Neural Plast. 2019 Jan 15;2019:2184398. doi: 10.1155/2019/2184398. PMID 30733800